CLINICAL TRIAL: NCT05828628
Title: A Prospective Imaging and Translational Tissue Study in CNS Lymphoma to Enable Further Disease Characterisation and the Development of Potential Predictive and Prognostic Biomarkers
Brief Title: CLIMB: CNS Lymphoma Imaging and Molecular Biomarkers Study
Acronym: CLIMB
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 5674
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-11

CONDITIONS: CNS Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine FFPE Tissue CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a new diagnosis of primary or secondary CNS lymphoma

SUMMARY:
A prospective imaging and translational tissue study in CNS lymphoma to enable further disease characterisation and the development of potential predictive and prognostic biomarkers.

DETAILED DESCRIPTION:
As a single centre exploratory study, this trial will recruit patients with newly diagnosed primary CNS lymphoma and will look at the molecular aspects of the disease in the tissue collection and imaging response assessments using CCA with respect to progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects capable of giving informed consent, or if appropriate, if subject's capacity is deemed limited due to CNS involvement, a consultee can provide consent on their behalf. Some patients with PCNSL may be incapable of providing their own consent due to the neurological effects of their disease. In these cases the patient will be classed as an incapacitated adult and a legal representative will be sought in accordance with English or Scottish law as applicable (see 7.2.1)
* A radiological or histological diagnosis of primary CNS lymphoma.
* Have not received prior CNS directed therapy. Prior use of steroids is permitted.
* Participants aged ≥18 years old.

Exclusion Criteria:

- Involvement of lymphoma outside of the CNS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed primary CNS lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Plasma ctDNA detection | 5 Years
  To assess if plasma ctDNA detection measured from end of treatment (using the tumour informed approach) can be used an early detection tool for progressive disease.
Contrast clearance analysis | 5 Years
  To assess the results of contrast clearance analysis

SECONDARY OUTCOMES:
Plasma ctDNA detection from end of treatment | 5 Years
  To assess if plasma ctDNA detection measured from end of treatment (using the tumour agnostic approach) can be used as an early detection tool for progressive disease
Plasma ctDNA detection rate at baseline | 5 Years
  To assess plasma ctDNA detection rate at baseline using the (i) tumour agnostic and (ii) tumour informed approach
Plasma ctDNA detection at end of treatment | 5 Years
  To assess whether plasma ctDNA detection at end of treatment can be used an early detection tool for progressive disease and survival using the (i) tumour agnostic and (ii) tumour informed approach
Plasma ctDNA detection rate at disease progression | 5 Years
  To assess plasma ctDNA detection rate at disease progression using the (i) tumour agnostic and (ii) tumour informed approach
Radiological data provided by CCA | 5 Years
  To evaluate whether additional radiological data provided by CCA is useful for prognostication and is associated with disease progression and survival

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chau, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Downs Road, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided